CLINICAL TRIAL: NCT00631098
Title: The Feasibility of Cannulating External Jugular Vein Compared With Cubital Vein (by Paramedics and Emergency Department Interns)
Brief Title: Cannulation for Resuscitation
Acronym: CARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Pasi Lahtinen, MD, Kuopio University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KUH5070198
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Resuscitation
Keywords: Resuscitation; venous cannulation; external jugular vein; cubital vein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cannulation of external jugular vein and cannulation of cubital vein
  Interventions: Procedure: venous cannulation

INTERVENTIONS:
Procedure: venous cannulation — External jugular and cubital vein cannulation

SUMMARY:
International CPR guidelines recommend the cannulation of a peripheral vein (antecubital or external jugular) during resuscitation. One reason for preferring the external jugular vein over more peripheral veins is the faster circulation time of drugs during CPR. The differences in circulation time may be over 90 seconds between peripheral and central (internal jugular) veins. However, cannulation of the external jugular vein may be more difficult and time consuming than cannulating cubital veins. There are no studies on the success rate, cannulation time and reliability of venous access comparing central and peripheral cannulation sites.

We hypothesized that cannulation of the external jugular vein (by paramedics and is a demanding procedure in an emergency situation and should not be recommended during resuscitation.

The aims of this study are to compare the feasibility of cannulating the external jugular vein compared to the cubital vein in terms of attempts, cannulation time and reliability of venous access.

DETAILED DESCRIPTION:
The protocol includes measurement of:

1. The time of cannulation
2. Number of attempts of cannulation, Every piercing of skin is counted as one attempt. Maximally three attempts will be allowed.
3. Failures. Perforation of vein and subcutaneous hemorrhage, arterial puncture, the appropriate vein is not found, free back flow of blood or free infusion of saline is not achieved the attempt are considered as failures . Cannulation of another site is then started or the study is ended.

The final protocol of the study will be a paired control, randomized prospective study. The randomization will be for the order of cannulation site (internal jugular or cubital vein first) In the final study the cannulation will be performed by emergency department interns and paramedics with advanced cardiac life support skills and licenced by Kuopio University Hospital.

For comparison and describing the experience of the paramedics an enquiry is accomplished and the following data are collected:

1. Age
2. Experience as a paramedic (years after graduation)
3. Theoretical guidance of cannulation (self estimated /hours)
4. Practical guidance of cannulation (self estimated/hours)
5. Experience of cannulation of the external jugular vein (self estimated/times)

For comparison and describing the experience of the interns in the ER a similar enquiry is accomplished,:

1. Age
2. Experience as an intern (years after graduation as MD)
3. Theoretical guidance of cannulation (self estimated /hours)
4. Practical guidance of cannulation (self estimated/hours)
5. Cannulation of external jugular vein (self estimated/times) Statistical analysis

The primary endpoint in this study is cannulation time of the two sites (internal jugular and cubital vein). The secondary end points are failure/success of cannulation and reliability of venous access as defined above.

Patient characteristics and anesthetic and operative variables are compared with the t-test for independent samples (continuous variables), or the Mann-Whitney U-test and 2-test (Pearson) or Fishers exact test when appropriate (categorical variables). Cannulation time differences between the groups will be compared with the t-test for independent samples (after tests for homoscedasticity and normality) or Mann-Whitney U-test if appropriate. Success of cannulation will be compared with 2-test (Pearson) or Fishers exact test when appropriate. A p value less than 0.05 is considered statistically significant. Results are given as mean (SD) or number of patients. All statistical analyses will be performed with SPSS version 11.01 software (SPSS Inc, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery patients

Exclusion Criteria:

* Morbid obesity (BMIover 35)
* Severe cardiac insufficiency (ejection fraction below 30%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure in this study is cannulation time of the two sites (internal jugular and cubital vein). | Cannulation time (minutes)

SECONDARY OUTCOMES:
The secondary end points are failure/success of cannulation and reliability of venous access. | success of cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Pasi K Lahtinen, MD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Department of Anesthesiology and Intensive Care/ Kuopio University hospital, Kuopio, Finland

REFERENCES:
- [Derived] Lahtinen P, Musialowicz T, Hyppola H, Kiviniemi V, Kurola J. Is external jugular vein cannulation feasible in emergency care? A randomised study in open heart surgery patients. Resuscitation. 2009 Dec;80(12):1361-4. doi: 10.1016/j.resuscitation.2009.08.026. Epub 2009 Oct 4. PMID 19804930